CLINICAL TRIAL: NCT06016439
Title: Outcomes of Different Treatment Modalities for Massive Rotator Cuff Tendon Tear.
Brief Title: Outcomes of Massive Rotator Cuff Tendon Tear Treatment.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tartu University Hospital (Other)
Collaborators: University of Tartu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tikk23
Record Dates: First submitted 2023-08-07; First posted 2023-08-29 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Syndrome
Keywords: rotator cuff injury; rotator cuff tears; massive; shoulder; shoulder injuries; superior capsular reconstruction; long head of biceps tendon; irreparable; tear; rupture; partial repair
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Injuries; Lacerations; Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arthroscopic rotator cuff partial repair with superior capsule augmentation with LHBBT (Experimental): If a tear is intra-operatively determined irreparable, randomization takes place.
  Irreparable tears that are randomly selected to receive arthroscopic rotator cuff partial repair including superior capsular augmentation with proximal part of the long head of the biceps tendon. The long head of the biceps tendon will be released from bicipital groove and proximal part of the tendon will be used to cover the rotator cuff gap and anchored to the greater tuberosity.
  Interventions: Procedure: Arthroscopic rotator cuff partial repair with superior capsular augmentation with LHBBT; Device: Suture anchor(s)
- Arthroscopic partial rotator cuff repair (Active Comparator): If a tear is intra-operatively determined irreparable, randomization takes place.
  Irreparable tears that are randomly selected to receive arthroscopic partial repair.
  Interventions: Procedure: Arthroscopic rotator cuff partial repair; Device: Suture anchor(s)
- Arthroscopic rotator cuff repair (Other): Arthroscopic complete repair.
  Interventions: Procedure: Arthroscopic complete rotator cuff repair; Device: Suture anchor(s)
- Rotator cuff tear conservative treatment (No Intervention): Conservative treatment following physiotherapy protocol.

INTERVENTIONS:
Procedure: Arthroscopic rotator cuff partial repair with superior capsular augmentation with LHBBT — Residual rotator cuff defect will be reconstructed using LHBBT.
  Arms: Arthroscopic rotator cuff partial repair with superior capsule augmentation with LHBBT
Procedure: Arthroscopic rotator cuff partial repair — Rotator cuff will be repaired with remaining residual defect.
  Arms: Arthroscopic partial rotator cuff repair
Procedure: Arthroscopic complete rotator cuff repair — Arthroscopic complete repair as a standard procedure.
  Arms: Arthroscopic rotator cuff repair
Device: Suture anchor(s) — Arthroscopic rotator cuff tendon(s) repair using suture anchor(s).
  Arms: Arthroscopic partial rotator cuff repair; Arthroscopic rotator cuff partial repair with superior capsule augmentation with LHBBT; Arthroscopic rotator cuff repair

SUMMARY:
Rotator cuff tear is the leading cause of shoulder pain in the elderly. There isn't enough evidence nor clinical guidelines to guide the treatment of massive rotator cuff tears, specially irreparable tears. Arthroscopic partial repair has been widely used and superior capsular reconstruction (SCR), either with allograft, autograft or augmentation with long head biceps brachii tendon (LHBBT), has been recently added. It is showing promising results, but lacking high quality evidence.

This is a prospective clinical study to compare the outcomes of different surgical methods for massive rotator cuff tendon tears. Minimal follow-up time will be two years. In this trial, massive rotator cuff tears will be anatomically repaired if possible. For irreparable tears a method will be randomly assigned intra-operatively once a tear is determined to be irreparable - either partial repair or partial repair with superior capsular reconstruction using the long head biceps brachii (LHBB) tendon. Patients who are eligible for the study but refuse operative treatment, will serve as conservative study group.

The hypothesis is that massive rotator cuff tears that are reparable will have the best functional outcomes. For irreparable tears, augmentation with LHBBT will give superior results over partial repair.

DETAILED DESCRIPTION:
Patients with massive rotator cuff tendon tears aged between 50 to 80 years will be included in the study following the eligibility criteria. Massive tear is defined as grade III tear according to Davidson and Burkhart classification (2010), supraspinatus (SSP) tendon retraction described by Patte (1990) classification.

The study is conducted in Tartu University Hospital Sports Traumatology Centre and rotator cuff repair procedures will be done by three orthopaedic surgeons with long experience in arthroscopic shoulder surgery.

It is determined intra-operatively whether the tear is reparable or not. If possible, the tendon(s) will be anatomically repaired. For irreparable tears intra-operative urn randomization takes place - either partial repair or partial repair with SCR using the LHBB tendon. Surgical techniques will be standardized. Patients who refuse operative treatment, will be followed as conservative treatment group.

The primary objective of the study is the functional status of the included subjects in different treatment groups. The secondary objective of the study is to confirm whether the tendons are intact on follow-up magnetic resonance imaging (MRI) 6 months, 12 months and 24 months after operation using Sugaya classification (2007).

The post-operative therapy regimen will be the same for each study group. Subjects will come for scheduled visits at 6-month, 12-month, and 24-month timepoints. Assessment tools consist of range of motion (ROM), strength measurements, preoperative radiography measuring acromio-humeral index (AHI), critical shoulder angle (CSA), acromion type and shoulder arthrosis (Hamada), functional scores: The Disabilities of the Arm, Shoulder and Hand (DASH), The Constant-Murley score (CMS), The American Shoulder and Elbow Surgeons (ASES) and visual analogue scale (VAS), also including Tampa kinesiophobia score and emotional well-being (EEK) score. Goutallier classification (1994) will be used pre- and postoperatively to measure muscle fatty infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Massive rotator cuff tendon tear: grade III according to Davidson and Burkhart 2010 classification, diagnosed on MRI, and LHBB tendon is intact.
* Primary rotator cuff pathology AND
* Symptoms have not lasted more than 6 months.
* In case of trauma, traumatic event no more than 6 months ago.
* Aged between 50 and 80 at the time of enrollment.
* Subject is able and willing to give informed consent AND
* Subject is physically and mentally willing and able to comply with the post-operative rehabilitation protocol, questionnaires, and scheduled clinical and radiographic visits.

Exclusion Criteria:

* Previous rotator cuff surgery of the index shoulder.
* Acute or chronic osteomyelitis.
* Inflammatory joint disease (rheumatoid arthritis/ (pseudo)gout arthritis).
* Uncontrolled diabetes.
* Active oncological disease.
* Radiologically stage IV shoulder joint arthrosis (rotator cuff arthropathy).
* Systemic or intra-articular corticosteroid therapy less than 60 days prior to planned operation date.
* Intramuscular or peroral corticosteroid treatment less than 30 days prior to planned operation date.
* Acute or chronic conditions that are contraindications for functional testing.
* MRI contraindicated.
* Substance or alcohol abuse.
* Refusal or withdrawal of consent.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2033-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Change in shoulder strength | Pre-operative baseline, 6-months, 12-months and 24-months follow-up visit
  Measured by the change in rotator cuff strength isokinetic testing (abduction, internal and external rotation).
Change in shoulder range of motion. | Pre-operative baseline, 6-months, 12-months and 24-months follow-up visit
  Measured by the change in shoulder range of motion (abduction, internal and external rotation).
Functional outcome according to the American Shoulder and Elbow Surgeons (ASES) score. | Pre-operative baseline, 6-months, 12-months and 24-months follow-up visit
  Measured by the change in joint functional score.
  The higher the score, the better the outcome.
  The patient self-assessment (pASES) includes 6 pain items and 10 functional items that are shoulder specific (Angst, 2008).
  The pASES form has 3 sections: pain, instability, activities of daily living (ADLs) (Goldhahn, 2008).
  Pain section: 4 questions with yes/no responses, 1 question covering number of pain tablets per day, and a VAS (visual analogue scale) from 0 (no pain) to 10 (worst pain).
  Instability section: 2 questions (1. Response yes/no about feelings of instability, 2. Quantify instability from 0 (stable) to 10 (very unstable)).
  Activities of daily living (ADLs): Each shoulder is included (affected/non affected), 10 items, with a 4 point ordinal scale, range: 0 (unable to perform activity) to 3 (no difficulty in doing activity) (Goldhahn 2008).
Functional outcome according to the Constant-Murley score (CMS). | Pre-operative baseline, 6-months, 12-months and 24-months follow-up visit
  Measured by the change in joint functional score.
  The higher the score, the higher the quality of the function.
  The test is divided into four subscales: pain (15 points), activities of daily living (ADL) (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points).
Functional outcome according to the Disabilities of the Arm, Shoulder and Hand (DASH). | Pre-operative baseline, 6-months, 12-months and 24-months follow-up visit
  Measured by the change in joint functional score.
  The higher the score, the more severe disability.
  30-item self-report questionnaire designed to assess symptoms and function of the entire upper extremity.
  Total scores range from 0 (minimum) to (100) maximum.
Change in pain score | Pre-operative baseline, 6-months, 12-months and 24-months follow-up visit
  Measured by the change in pain score according to the visual analogue scale (VAS) from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Integrity of surgically repaired rotator cuff tendons on MRI studies using Sugaya classification (2005). | postoperatively 6 months, 12 months and 24 months
  Integrity of surgically repaired rotator cuff tendons on post-operative MRI studies.
  Classified into five categories (from intact tendon to full tear):
  Type I: sufficient thickness with homogeneously low intensity; Type II: sufficient thickness with partial high intensity; Type III: insufficient thickness without discontinuity; Type IV: the presence of a minor discontinuity; Type V: the presence of a major discontinuity.
Change in quality of life | Pre-operative baseline, 6-months, 12-months and 24-months follow-up visit
  Measured by the change in score according to EEK-2 (emotsionaalse enesetunde küsimustik, Emotional State Questionnaire) score.
  The higher the score, the higher the risk of having emotional state disabilities.
  The overall score ranges from 0-112, but it is divided into six categories that are assessed separately.
Change in kinesiophobia score | Pre-operative baseline, 6-months, 12-months and 24-months follow-up visit
  Change in kinesiophobia score according to Tampa Scale for Kinesiophobia.
  The higher the score, the higher the degree of kinesiophobia.
  Results consist of a total raw score (range between 17 and 68) and two subscale scores (activity avoidance and somatic focus).

CONTACTS AND LOCATIONS:
Overall Officials: Tiina Tikk, MD, Principal Investigator — University of Tartu

IPD SHARING:
Plan to Share IPD: No